CLINICAL TRIAL: NCT02834871
Title: Integration of the Cervical Proprioceptive Signals in Patients With Cervical Dystonia
Acronym: STAC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SSA_2014_23
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with cervical dystonia (Other): Computerized assessment of the cervical muscular force and with electromyogram in patients with cervical dystonia
  Interventions: Device: Electromyogram
- patients without cervical dystonia (Other): Computerized assessment of the cervical muscular force and with electromyogram in patients without cervical dystonia
  Interventions: Device: Electromyogram

INTERVENTIONS:
Device: Electromyogram

SUMMARY:
The purpose of this study is to compare the cervical muscular force control , taking into account the proprioceptive signals, in patients with and without cervical dystonia.

ELIGIBILITY:
Inclusion criteria:

* patients presenting focal or segmental cervical dystonia diagnosed by a neurologist expert in the diseases with abnormal movements
* having signed a consent for study participation

No Inclusion Criteria:

Neurological affection other than cervical dystonia (typical or atypical parkinsonism, other ...)

* Severe pain, trauma or disease of the cervical spine known or suspected other than cervical dystonia requiring treatment in the last 6 months
* Ongoing neuroleptic treatment
* Pregnancy or breastfeeding
* Lack of insurance coverage

For patients, are added the following no inclusion criteria are added:

* Trembling cervical dystonia
* Injection of botulinum toxin in the past three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Measuring (in Newton) of the muscular force exerted by extending movements of the cervical spine in static and dynamic condition | two hours

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmique Adolphe de Rothschild, Paris, Paris, France

REFERENCES:
- [Result] Carment L, Maier MA, Sangla S, Guiraud V, Mesure S, Vidailhet M, Lindberg PG, Bleton JP. Does dystonic muscle activity affect sense of effort in cervical dystonia? PLoS One. 2017 Feb 13;12(2):e0172019. doi: 10.1371/journal.pone.0172019. eCollection 2017. PMID 28192488